CLINICAL TRIAL: NCT01728948
Title: Non-interventional Study of Effectiveness of Elderly Metastatic Renal Cell Carcinoma (mRCC) Treated With Sorafenib
Brief Title: Sorafenib in Elderly mRCC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16399; NX1212CN (Other: company internal)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Sorafenib; renal cell carcinoma(RCC); elderly; effectiveness; safety
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — treatment (including dose, duration, modification) decided by the investigator

SUMMARY:
This prospective, single arm, multi-center pilot study includes 120 mRCC patients over 65 years, no prior systemic treatment, determined to be candidates for systemic therapy by the investigator. The treatment with Sorafenib should comply with the recommendations written in the local product information. The primary endpoint is overall survival. The secondary endpoints including other effectiveness points, safety and patients characteristics. With 120 completed patients, if the observed survival rate at 12 months is 60%, the width of a 95% confidence interval will be approximately 18%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically/cytologically diagnosed metastasis RCC who are candidates for systemic therapy and have decided to accept Sorafenib treatment.
* >=65 years of age
* Patients who have signed the informed consent
* Patients with a life expectancy of ≥12 weeks
* No prior systemic treatment

Exclusion Criteria:

* The approved local product label must be followed for the exclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: mRCC patients, >= 65 years of age, No prior systemic treatment, need systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01-06 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 2.5 years

SECONDARY OUTCOMES:
Progression free survival by the Response Evaluation Criteria in Solid Tumor (RECIST) Criteria | up to 2.5 years
Disease control rate by the Response Evaluation Criteria in Solid Tumor (RECIST) Criteria | up to 2.5 years
Survival rate by one year | up to 1 year
Number of participants with adverse events (AE) and Serious adverse events (SAE) as a measure of safety and tolerability | up to 3.5 years
Patient characteristics (birthdate (at least year), sex, weight, height, etc) | up to 2.5 years
Response rate (RR) | up to 3.5 years
Time to first relief of clinical symptoms and physical signs | up to 3.5 years
Treatment pattern | up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China